CLINICAL TRIAL: NCT05117268
Title: ASSESSMENT OF SDF vs. GIC AND HALL TECHNIQUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUI/CTR/2021/7
Record Dates: First submitted 2021-11-04; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A facial image scale shall be shown to participants before treatment and immediately after treatment to determine child anxiety with each treatment where the child will be asked to identify the face that best expressed their feeling at that point of time.
  Possible adverse events of each treatment shall be recorded by registering any complaint of sensitivity, gingival irritation, tattoo formation, burning, unpleasant taste, silver allergy and nausea. To assess parental aesthetic perception, a questionnaire will be presented that specifically asks if they were annoyed by the appearance of their child, or the child avoided smiling.
Masking Description: No masking strategy is selected because intervention to be performed in all 3 groups is different. Operator cannot be blinded. Consent is necessary for SDF application. For the reasons listed, patient cannot be blinded for the procedure to be done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silver Diamine Fluoride (Experimental): In the experimental group, 44 children will be provided with SDF application, after gross debris removal to allow better contact of SDF. The entire dentition will be treated with sodium chloride fluoride varnish to prevent caries.
  Interventions: Procedure: SDF Application for caries arrest
- Glass Ionomer Restoration (Placebo Comparator): In placebo control group n= 44 participants will be enrolled. High viscosity glass ionomer restoration will be placed after complete caries excavation using high-speed handpiece and air/water coolant. Patient will be dispensed with clear postoperative instructions.
  Interventions: Procedure: Glass ionomer restoration
- Hall Technique (Active Comparator): In active comparator group, n= 44 study participants will be enrolled. Pre-formed metal crowns will be selected according to the tooth size and filled with low viscosity glass ionomer cement and seated using digital/ finger pressure.
  Interventions: Procedure: Hall technique

INTERVENTIONS:
Procedure: SDF Application for caries arrest — Intervention will be performed by trained consultants following the recommended protocol for SDF application: (A) Gross debris will be removed from cavity to allow better contact with SDF; (B) Protective coating of petroleum jelly will be applied to surrounding facial skin and lips to prevent chances of temporary tattoo formation; (C) Area to be treated shall be isolated using cotton rolls and saliva ejectors to prevent gingival irritation; (D) Extra caution will be exercised when applying SDF on primary teeth adjacent to permanent teeth to avoid inadvertent black staining; (E) One drop will be used used for the whole appointment. Bent micro-brush is to be used for application time of 1 min is to be used to reduce systemic absorption; (F) Compressed air shall be applied with gentle flow for up to 3 minutes. Entire dentition will be treated with sodium fluoride varnish to prevent caries
  Arms: Silver Diamine Fluoride
Procedure: Glass ionomer restoration — The lesions of control group glass ionomer restoration group will be treated according to following clinical protocol: (A) Isolation of treatment area using cotton rolls and saliva ejectors; (B) Carious lesion excavation using high speed handpiece; (C) High viscosity glass ionomer cement mixed following manufacturer's instructions; (D) Cavity will be slightly overfilled using a flat plastic instrument, the occlusal surface will be protected with Vaseline and gloved finger will be used to apply slight pressure for 30s. Postoperative instructions will be clearly explained to each patient caregiver.
  Arms: Glass Ionomer Restoration
Procedure: Hall technique — In Hall technique, correct size preformed metal crown will be selected and shall be placed without caries excavation. The crown will be filled with glass ionomer cement and seated with finger pressure. Local anesthesia was not used finger pressure was maintained on the crown until the glass ionomer cement was set.
  Arms: Hall Technique

SUMMARY:
Early childhood caries (ECC) ,a global public health problem, highly prevalent and severe with life long implications is entirely preventable.

as an alternative to general anesthesia low cost innovative materials such as SDF are promising for low income countries such as Pakistan for reducing the burden of dental caries.

SDF may positively transform prevntive and clinical pediatric dental practices and services in Pakistan.

FDA approves 38% SDF for arresting caries in vulnerable populations.

DETAILED DESCRIPTION:
The study will be conducted at Pediatric Dentistry Department of Foundation University College of Dentistry and Hospital. Participants (beneficiary entitled patients consenting for treatment) will be enrolled from patients looking for dental treatment at outpatient pediatric dentistry clinic. Written and verbal informed consent will be taken from each patient guardian. Aims and objectives of study will be clearly explained to participants. Confidentiality will be maintained throughout the study length and right to withdraw from the study will be warranted to all participants. Children will be recruited applying following selection criteria mentioned. Baseline information, like previous dental experience, history of carbonated drinks and dietary sugar intake, experience with local anesthesia, parental education status and socioeconomic status will be recorded. Detailed intra-oral examination will be carried out using mouth mirror, dental probe and triple syringe. Cavitated lesions will be assessed and receive ICDAS score. Cavities with ICDAS code 4, 5 and 6 are to be enrolled in the study. In SDF group, informed consent will be taken from parents, clearly explaining the potential for black staining. Intervention will be performed by trained consultants following the recommended protocol for SDF application: (A) Gross debris will be removed from cavity to allow better contact with SDF; (B) Protective coating of petroleum jelly will be applied to surrounding facial skin and lips to prevent chances of temporary tattoo formation; (C) Area to be treated shall be isolated using cotton rolls and saliva ejectors to prevent gingival irritation; (D) Extra caution will be exercised when applying SDF on primary teeth adjacent to permanent teeth to avoid inadvertent black staining; (E) One drop will be used used for the whole appointment. Bent micro-brush is to be used for application time of 1 min is to be used to reduce systemic absorption; (F) Compressed air shall be applied with gentle flow for up to 3 minutes. Entire dentition will be treated with sodium fluoride varnish to prevent caries.

The lesions of control group glass ionomer restoration group will be treated according to following clinical protocol: (A) Isolation of treatment area using cotton rolls and saliva ejectors; (B) Carious lesion excavation using high speed handpiece; (C) High viscosity glass ionomer cement mixed following manufacturer's instructions; (D) Cavity will be slightly overfilled using a flat plastic instrument, the occlusal surface will be protected with Vaseline and gloved finger will be used to apply slight pressure for 30s. Postoperative instructions will be clearly explained to each patient caregiver. In Hall technique, correct size preformed metal crown will be selected and shall be placed without caries excavation. The crown will be filled with glass ionomer cement and seated with finger pressure. Local anesthesia was not used finger pressure was maintained on the crown until the glass ionomer cement was set.

Primary outcome was caries-arresting potential of all three treatment groups. Recall examination was performed at 6 and 12 months. At each recall, ICDAS scores were compared to initial values of teeth. Treatment was classified as success when caries on teeth was classified as inactive based on lower ICDAS score compared to initial scores. Treatment was considered a failure if lesion had progressed to higher score at review examination. Presence of spontaneous pain, sensitivity to percussion and periapical swelling was also considered a failure. Visual and tactile examination was also done to check if the lesion was hard on gentle probing. Secondary outcome was parental aesthetic perception. Factors such as child anxiety, treatment time, adverse events like gingival irritation, burning of mucosa and bad taste, were all taken into account.

A facial image scale was shown to participants before treatment and immediately after treatment to determine the level of child's anxiety with each treatment. Child patient was asked to select from series of facial expressions (very happy, happy, neutral, unhappy, and very unhappy), the face that best expressed their feeling at that point in time. Time required for each treatment group was calculated using a digital timer. Possible adverse events of each treatment were recorded. Any complaint of sensitivity, gingival irritation, tattoo formation, burning, unpleasant taste, silver allergy and nausea was registered immediately. To assess parental aesthetic perception, they were asked questions like if they were displeased by the appearance of their child, or if the child avoided smiling.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders.
* Age range between 5 to 10 years old.
* Both deciduous maxillary and mandibular untreated teeth.
* Carious teeth categorized as ICDAS code 4, 5 and 6 will be included.
* Active carious lesions on occlusal surface of primary molars

Exclusion Criteria:

Permanent dentition will be excluded from this study

* Primary molar showing signs of irreversible pulpitis
* Patients diagnosed with periapical abscess
* Patients allergic to silver
* Medically compromised or patients with childhood impairment and disability.
* Hemophilic patients
* Epileptic patients
* Non-consenting patients for silver staining

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Caries arresting potential of all 3 treatment groups | 6 months
  At each recall, ICDAS scores were compared to initial values of teeth. Treatment was classified as success when caries on teeth was classified as inactive based on lower ICDAS score compared to initial scores

SECONDARY OUTCOMES:
Parental aesthetic perception questionnaire. | 24 hours
Facial Image scale for child anxiety | 24 hours
Treatment time through digital timer | 24 hours
Gingival irritation from follow-up interview | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No